CLINICAL TRIAL: NCT06834659
Title: CRANIUM: Post-Market Performance Follow-up Study for the Evaluation of the Presence of Circulating Plasma Brain Biomarkers in Peripheral Blood and Acute Traumatic Brain Injury in Adult Emergency Department Patients.
Brief Title: Correlation and Rapid Analysis of Neurological Injury Using Markers
Status: Not yet recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Di Resta, PhD, Università Vita-Salute San Raffaele
Other Study IDs: CRANIUM
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury (TBI) Patients
Keywords: Biomarkers; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with TBI: Adult patients (ages ≥18 and ≤65), conscious and unconscious, presenting to the emergency department with TBI at triage. TBI is defined as trauma caused by an external physical force capable of causing temporary or permanent alterations in consciousness and/or neurological function.
  Post Market Performance follow-up study: Application of the Abbott i-STAT™ TBI Plasma Test to all cases within 12 hours of cranial trauma for detecting GFAP and UCH-L1 biomarkers.

SUMMARY:
Each year, approximately 69 million people worldwide suffer from traumatic brain injuries (TBI), representing a significant burden on public health, society, and the economy. Timely and accurate care can influence short-, medium-, and long-term outcomes, making the reduction of diagnostic delays crucial. TBI diagnostics require careful consideration, as initial evaluations may differ from final assessments, and patient conditions may evolve over time.

In this monocentric, observational, post-market follow-up study we aim to evaluate the Abbott i-STAT™ TBI Plasma Test in detecting circulating brain biomarkers (GFAP and UCH-L1) in adult patients with TBI.

The study involves recruiting 200 adult patients (aged 18-65 years) presenting to the emergency department with TBI over a two-year period. For each participant, a blood sample will be collected as part of routine clinical care and analyzed using the Abbott i-STAT™ TBI Plasma Test within 12 hours of the trauma. The results will be compared with those obtained from cranial CT scans, the gold standard for diagnosing intracranial injuries.

Specifically, the study aims to assess the diagnostic accuracy of the test in excluding intracranial injuries, particularly in cases of mild TBI, and to explore potential correlations between biomarker presence and injury severity. No additional procedures beyond routine clinical care are required, and all collected data will be used exclusively for the study's predefined objectives.

DETAILED DESCRIPTION:
Post-Market Performance Follow-up Study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65, male and female, presenting to the emergency department due to TBI, defined as trauma caused by an external force leading to temporary or permanent alterations in consciousness and/or neurological function. TBI severity is evaluated using the Glasgow Coma Scale (GCS).
* Sign of informed consent by patient or legal tutor

Exclusion Criteria:

* Pediatric patients (<18 years).
* Patients >65 years, to avoid potential confounding factors such as elevated GFAP levels associated with Alzheimer's disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adult patients aged between 18 and 65 years, conscious and unconscious, who present to the emergency department with traumatic brain injury (TBI) at triage. TBI is defined as trauma resulting from an external physical force capable of causing temporary or permanent alterations in consciousness and/or neurological function. The clinical severity of TBI (mild, moderate, or severe) will be assessed using the Glasgow Coma Scale (GCS), ensuring alignment with the study objectives.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the real-world effectiveness of the innovative technology | T1: first blood sample for biomarker testing and CT scan within 12 hours of trauma; T2: second blood sample for biomarker testing and CT scan at 12 to 24 hours post-initial evaluation, if clinically indicated due to neurological deterioration.
  Concordance Between Abbott i-STAT™ TBI Plasma Test Results and Cranial CT Scan in mTBI Cases.
  The primary outcome measure is the percentage agreement between the qualitative result of the Abbott i-STAT™ TBI Plasma Test (positive or negative) and the presence or absence of traumatic brain injury (TBI) or intracranial haemorrhages detected by cranial CT scan in patients with mild traumatic brain injury (mTBI).

OTHER OUTCOMES:
Exploring the correlation between a positive result from the Abbott test and the progression of intracranial injuries (ICI) detected via CT scan, specifically in patients for whom a second CT scan is deemed necessary and performed. | T1: first blood sample for biomarker testing and CT scan within 12 hours of trauma; T2: second blood sample for biomarker testing and CT scan at 12 to 24 hours post-initial evaluation, in cases with neurological deterioration.
  The study will evaluate potential relationships between biomarkers identified by the test and the severity of the intracranial damage.
  This approach will allow for a comparative analysis of the presence of biomarkers in the peripheral blood and their association with evolving intracranial conditions. The study seeks to validate the clinical relevance of biomarkers in predicting not only the presence but also the extent and progression of intracranial damage.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oris C, Bouillon-Minois JB, Kahouadji S, Pereira B, Dhaiby G, Defrance VB, Durif J, Schmidt J, Moustafa F, Bouvier D, Sapin V. S100B vs. "GFAP and UCH-L1" assays in the management of mTBI patients. Clin Chem Lab Med. 2023 Dec 1;62(5):891-899. doi: 10.1515/cclm-2023-1238. Print 2024 Apr 25. PMID 38033294